CLINICAL TRIAL: NCT03054324
Title: FFRB Study: Validation of a Predictive Model of Coronary Fractional Flow Reserve in Patients With Intermediate Coronary Stenosis
Brief Title: Validation of a Predictive Model of Coronary Fractional Flow Reserve in Patients With Intermediate Coronary Stenosis
Acronym: FFRB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/2097
Record Dates: First submitted 2017-02-06; First posted 2017-02-15 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-03

CONDITIONS: Coronary Stenosis
Keywords: Cardiovascular Diseases; Fractional Flow Reserve; Ischemic Heart Disease; CT Angiogram
MeSH Terms: conditions — Coronary Stenosis; Cardiovascular Diseases; Myocardial Ischemia | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fractional Flow Reserve — Coronary fraction flow reserve (FFR), the ratio of the mean coronary pressure distal to a coronary stenosis to the mean aortic pressure during maximal coronary blood flow (hyperemia), defines the hemodynamic significance of coronary artery narrowing.

SUMMARY:
Coronary fraction flow reserve (FFR), the ratio of the mean coronary pressure distal to a coronary stenosis to the mean aortic pressure during maximal coronary blood flow (hyperemia), defines the hemodynamic significance of coronary artery narrowing. Noninvasive assessment of FFR via a combination of computational fluid dynamics (CFD) and coronary CT angiography CCTA (the so-called FFRCT) has potential. Coronary computed tomographic angiography is a noninvasive test for diagnosis of anatomic coronary stenosis (i.e., narrowing of a blood vessel). A new analytical model of FFR from the general Bernoulli equation (conservation of energy) (FFRB) is simple and has potential. A collaborator group has recently developed a new analytical model to quantify pressure drop, and hence FFR, based on lesion dimensions (i.e., the cross-section area along the lesion and the length of lesion) and coronary flow, with no empirical parameters. The investigators hypothesize that this new model will allow quantification of FFR (FFRB) in a cohort of human patients with intermediate coronary stenosis. The study will compare FFRB with invasive FFR measurements from invasive coronary angiography (ICAG).

DETAILED DESCRIPTION:
Coronary fraction flow reserve (FFR), the ratio of the mean coronary pressure distal to a coronary stenosis to the mean aortic pressure during maximal coronary blood flow (hyperemia), defines the hemodynamic significance of coronary artery narrowing. Recent landmark studies showed a clear benefit of FFR in guiding percutaneous coronary intervention (PCI) for better clinical outcome and cost-effectiveness. The reference method for FFR measurement requires the use of a pressure wire inserted across the stenosis invasively. Therefore, a non-invasive method to quantify FFR is clinically desired.

Noninvasive assessment of FFR via a combination of computational fluid dynamics (CFD) and coronary CT angiography CCTA (the so-called FFRCT) has potential. Coronary computed tomographic angiography is a noninvasive test for diagnosis of anatomic coronary stenosis (i.e., narrowing of a blood vessel). However, CCTA alone does not determine whether a stenosis causes ischemia. Computational fluid dynamics (CFD), applied to CCTA images, enables computation of FFR (FFRCT). Recent studies have demonstrated the potential of FFRCT as a promising noninvasive method for identification of individual lesion with ischemia from both single centre and multi-centre prospective studies. However, the FFRCT is currently performed remotely and it takes several hours to complete the computation for each study. This potentially impedes the wider clinical application of FFRCT.

A new analytical model of FFR from the general Bernoulli equation (conservation of energy) (FFRB) is simple and has potential. The Bernoulli equation has many clinical applications. A collaborator group has recently developed a new analytical model to quantify pressure drop, and hence FFR, based on lesion dimensions (i.e., the cross-section area along the lesion and the length of lesion) and coronary flow, with no empirical parameters. The investigators validated it using in vitro and in vivo experiments and finite-element method. The study team hypothesize that this new model will allow quantification of FFR (FFRB) in a cohort of human patients with intermediate coronary stenosis. The investigators will compare FFRB with invasive FFR measurements from invasive coronary angiography (ICAG).

Aims and Objectives

Primary aim: Diagnostic performance of FFRB with CCTA data in patients with intermediate coronary artery disease (CAD), as compared to an invasive FFR reference standard (FFR<=0.80)

Secondary aims: Diagnostic performance with FFRB for lesions of intermediate stenosis severity; Determining the per-vessel correlation of FFRB value to FFR from ICA

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-98.
* Underwent CCTA within 180 days and is scheduled to undergo coronary angiography and FFR in vessels having diameter stenosis between 30-90%, and deemed clinically indicated for evaluation.

Exclusion Criteria:

* Previous PCI
* Previous coronary artery bypass surgery
* Contraindication to beta blockers , nitroglycerin or adenosine, including second- or third-degree heart block; sick sinus syndrome; long QT syndrome; severe hypotension; asthma, chronic obstructive pulmonary disease, heart rate <50 beats/min.
* Acute coronary syndrome (acute myocardial infarction, unstable angina or unstable arrhythmias) is suspected.
* Had recent myocardial infarction within 30 days before CCTA or between CCTA and coronary angiography
* Has known complex congenital heart disease.
* Has had pacemaker or internal defibrillator leads implanted.
* Has a prosthetic heart valve or significant valvular pathology.
* Has tachycardia or significant arrhythmia; heart rate ≥ 100 beats/min; systolic blood pressure ≤90 mmHg.
* Renal dysfunction (glomerular filtration rate (GFR) <30 mL/min/1.73m2).
* Allergy to iodinated contrast.
* Individuals unable to provide informed consent.
* Non-cardiac illness with life expectancy <2 years.
* Pregnant state.
* Canadian Cardiovascular Society class IV angina.
* Patients with a left ventricular ejection fraction less than 30%.
* Patients with hypertrophic cardiomyopathy.

Ages: 21 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 132 patients scheduled to undergo clinically indicated invasive coronary angiography (ICAG) and who had CCTA performed within 180 days before the scheduled ICA, will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2016-09-02 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of FFRB to invasive FFR | 6 months from CT Angiogram
  The diagnostic performance of FFRB with CCTA data in patients with intermediate coronary artery disease (CAD), as compared to an invasive FFR reference standard (FFR<=0.80)

SECONDARY OUTCOMES:
Diagnostic performance with FFRB for lesions of intermediate stenosis severity | 6 months from CT Angiogram
Per-vessel correlation of FFRB to invasive FFR | 6 months from CT Angiogram

CONTACTS AND LOCATIONS:
Overall Officials: Soo Teik Lim, MBBS, Principal Investigator — National Heart Centre Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - National Heart Centre Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang C, Leng S, Tan RS, Chai P, Fam JM, Teo LLS, Chin CY, Ong CC, Baskaran L, Keng YJF, Low AFH, Chan MY, Wong ASL, Chua SJT, Wu Q, Tan SY, Lim ST, Zhong L. Coronary CT Angiography-based Morphologic Index for Predicting Hemodynamically Significant Coronary Stenosis. Radiol Cardiothorac Imaging. 2023 Dec;5(6):e230064. doi: 10.1148/ryct.230064. PMID 38166346